CLINICAL TRIAL: NCT02844270
Title: The Feasibility, Safety and Efficacy Evaluation of Galaxy Rapamycin Drug-Eluting Bioresorbable Coronary Stent System for the Treatment of Coronary Heart Disease: a First-in-man Study
Brief Title: Galaxy Rapamycin Drug-Eluting Bioresorbable Coronary Stent System First-in-man Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Bio-heart Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALAXY-2015-01
Record Dates: First submitted 2016-07-13; First posted 2016-07-26 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galaxy stent (Experimental): The galaxy Rapamycin Drug-Eluting Bioresorbable Coronary Stent System will be implanted in all subjects.
  Interventions: Device: Rapamycin Drug-Eluting Bioresorbable Coronary Stent System

INTERVENTIONS:
Device: Rapamycin Drug-Eluting Bioresorbable Coronary Stent System — Implantation of the Rapamycin Drug-Eluting Bioresorbable Coronary Stent System
  Other Names: Galaxy

SUMMARY:
The Galaxy First-in-man study is a small pilot. single arm research , which will enroll a total of 45 patients. The goal is to access the feasibility, safety and efficacy of Rapamycin Drug-Eluting Bioresorbable Coronary Stent System in the treatment of patients with de novo coronary lesion.

DETAILED DESCRIPTION:
This study is a prospective, single arm clinical trial. 45 patients enrolled in the study will be randomly assigned to queue1 (n=30) and queue 2 (n=15). The clinical follow-up will be performed in all subjects at 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after stent implantation; angiographic,IVUS and OCT follow-up will be performed at 6 months and 2 years after stent implantation in queue 1; angiographic,IVUS and OCT follow-up will be performed at 1 year and 3 years after stent implantation in queue 2. The primary endpoint of the study is target lesion failure (TLF) at 30 days after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age, males or non-pregnant females;
* With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction;
* Total number of target lesion is 1;
* Target lesion must be ≤ 25mm in length (visual estimation) and 3.0 to 3.75 mm in diameter ;
* Visual assessment of target lesion diameter stenosis ≥ 70%,TIMI blood flow≥1;
* The target lesion can be covered by one stent;
* Patient must be an acceptable candidate for coronary artery bypass graft;
* To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

* Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
* Implantation of stent in target vessel within 1 year , patients with planned intervention again within six months;
* Severe congestive heart failure (NYHA class III and above) ,left ventricular ejection fraction or <40% (ultrasound or left ventricular angiography);
* Preoperative renal function serum creatinine >2.0mg/DL; receiving hemodialysis;
* Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
* Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
* The patient's life expectancy is less than 12 months;
* To participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
* Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
* Heart transplantation patients;
* The unstable arrhythmia, such as high risk ventricular extrasystole and ventricular tachycardia;
* Cancer need chemotherapy;
* Immunosuppression and autoimmune diseases, planned or undergoing immunosuppressive therapy;
* Planning or being receiving long-term anticoagulant therapy, such as heparin, warfarin, etc;
* Within six months for elective surgery requires stopping aspirin, Clopidogrel patients;
* Blood test prompted platelet counts of less than 100x10E9/L or greater than 700x10E9/L, white blood cells than 3x10E9/L; known or suspected liver disease (such as hepatitis);
* Peripheral vascular disease, 6F catheter is not available.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-08-09 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Device-related composite endpoints (Target Lesion Failure) | 1 month after stent implantation
  contains cardiac death,target vessel myocardial infarction and clinical driven-target lesion revascularization

SECONDARY OUTCOMES:
Device Success | From the start of index procedure to end of index procedure
  Successful delivery and deployment of the assigned stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-stent residual stenosis of less than 30% by quantitative coronary angiography (QCA)
Procedural Success | At time of procedure up to 7 days in hospital
  Achievement of final in-stent residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one assigned stent at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR.
Target Lesion Failure | 6 months
  Target lesion failure is a composite endpoint of cardiac death, target vessel related myocardial infarction (TV-MI) and the ischemia-driven target lesion revascularization
Target Lesion Failure | 1 year
Target Lesion Failure | 2 years
Target Lesion Failure | 3 years
Target Lesion Failure | 4 years
Target Lesion Failure | 5 years
Patient Oriented Composite Endpoint | 30 days
  Patients oriented composite endpoint includes all-cause death, all myocardial infarction and any revascularization
Patient Oriented Composite Endpoint | 6 months
Patient Oriented Composite Endpoint | 1 year
Patient Oriented Composite Endpoint | 2 years
Patient Oriented Composite Endpoint | 3 years
Patient Oriented Composite Endpoint | 4 years
Patient Oriented Composite Endpoint | 5 years
Stent Thrombosis | 30 days
Stent Thrombosis | 6 months
Stent Thrombosis | 1 year
Stent Thrombosis | 2 years
Stent Thrombosis | 3 years
Stent Thrombosis | 4 years
Stent Thrombosis | 5 years
Minimal lumen diameter | 6 months, 1year, 2 years and 3years
In-stent stenosis | 6 months, 1year, 2 years and 3years
Late lumen loss | 6 months, 1year, 2 years and 3years
Covered struts percentage | 6 months, 1year, 2 years and 3years
Malapposed struts percentage | 6 months, 1year, 2 years and 3years
Neointimal hyperplasia area | 6 months, 1year, 2 years and 3years
Neointimal hyperplasia area obstruction | 6 months, 1year, 2 years and 3years
Struts core area | 6 months, 1year, 2 years and 3years
Struts neointimal thickness | 6 months, 1year, 2 years and 3years
IVUS mean vessel area | 6 months, 1year, 2 years and 3years
IVUS mean lumen area | 6 months, 1year, 2 years and 3years
IVUS mean strut area | 6 months, 1year, 2 years and 3years

IPD SHARING:
Plan to Share IPD: Undecided